CLINICAL TRIAL: NCT05911425
Title: Envolizumab in Combination With Sovalteinib for the Treatment of Treated Bile Duct Cancer in an Open, Single-arm, Phase II Clinical Study
Brief Title: Combined Treatment of Treated Bile Duct Cancer
Acronym: CHOL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Luo Cong, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-222
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bile Duct Cancer
MeSH Terms: conditions — Bile Duct Neoplasms

STUDY DESIGN:
Intervention Model Description: envolizumab sovalteinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective Research (Other): Envolizumab 300mg, Q2W, day 1, subcutaneous injection Soventinib 200mg, Q2W, once daily, orally Every 2 weeks as a cycle.
  Interventions: Drug: envolizumab , sovalteinib

INTERVENTIONS:
Drug: envolizumab , sovalteinib — Envolizumab 300mg, Q2W, day 1, subcutaneous injection Soventinib 200mg, Q2W, once daily, orally Every 2 weeks as a cycle.

SUMMARY:
The study will evaluate the efficacy and safety of envelizumab in combination with sovalteinib in the treatment of treated bile duct cancer, and explore treatment options to improve patient survival, while the study will attempt to explore the characteristics of the population benefiting from the treatment, and construct a preliminary efficacy prediction model by detecting markers in blood to provide a theoretical basis for implementing precise treatment.

ELIGIBILITY:
Inclusion Criteria:

1. the patient is 18-75 years old, can fully understand the content of this study, voluntarily join this study and cooperate with the study, and has full civil capacity
2. have a histologically or cytologically confirmed diagnosis of bile duct cancer
3. Patients with cholangiocarcinoma who have previously failed (disease progression or intolerability) to receive first-line or higher standard-containing therapy, including but not limited to chemotherapy, immunotherapy, targeted therapy, etc.; or who have relapsed within 6 months of postoperative adjuvant therapy;
4. patients receiving the first dose of this study at an interval of ≥ 28 days from the last treatment;
5. having a measurable lesion (≥10 mm long diameter on CT scan for non-lymph node lesions and ≥15 mm short diameter on CT scan for lymph node lesions according to RECIST 1.1 criteria)
6. an ECOG PS score: 0 to 1;
7. subjects voluntarily enrolled in this study, with good compliance and cooperation with safety and survival follow-up.
8. have adequate organ function and have not had a blood transfusion, used granulocyte colony-stimulating factor (G-CSF), or used medication within 7 days prior to screening to correct: 1) Blood count: Absolute Neutrophil Count (ANC) 1.5 × 109/L, Platelet (PLT) ≥ 70 × 109/L, Hemoglobin (HGB) ≥ 90 g/L; 2) Liver function: serum total bilirubin (Total Bilirubin, TBIL) ≤ 1.5 × Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤3×ULN; serum albumin ≥28 g/L; Alkaline Phosphatase (ALP) ≤5×ULN; after conventional hepatoprotective treatment meeting the above criteria, and can be stable for at least 1 week after evaluation by the investigator can be enrolled; 3) Renal function: serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/mi (applying the standard Cockcroft-Gault formula); (4) Coagulation: International Normalized Ratio (INR) ≤ 1.5 /PT ≤ 1.5 × ULN, aPTT ≤ 1.5 × ULN; (5) nutritional status: body mass index BMI ≥ 18 kg/m2, weight ≥ 40 kg, serum albumin ≥ 3.0 g/dL;
9. life expectancy ≥ 6 months.

Exclusion Criteria:

1. subjects with prior or concurrent other malignancies, including combined or mixed hepatocellular/cholangiocarcinoma or potbelly cancer;
2. active brain metastases or spinal cord compression;
3. not having received systemic antitumor therapy prior to the first study drug treatment
4. prior antitumor therapy-related toxicity not recovered to CTCAE ≤ grade 1, except for alopecia and platinum-induced peripheral neuropathy ≤ grade 2
5. prior liver transplantation;
6. the subject has known prior hypersensitivity to macromolecular protein agents or drug components of sovalteinib
7. subject has any active autoimmune disease or history of autoimmune disease (e.g., the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, previous thyroid surgery cannot be included; subject has vitiligo or asthma that has completely resolved in childhood and does not require any intervention in adulthood (subjects with vitiligo or asthma that has been in complete remission in childhood and does not require any intervention as an adult may be included; subjects with asthma requiring medical intervention with bronchodilators are not included);
8. subjects who are on immunosuppressive, immunomodulatory, or systemic, or absorbable topical hormone therapy for immunosuppressive purposes (doses >10 mg/day of prednisone or other equipotent hormone) and who continue to use them within 2 weeks prior to enrollment
9. clinically symptomatic ascites or pleural effusion that is not controlled by medication and requires therapeutic puncture or drainage prior to the first study drug therapy;
10. have had major surgical procedures or surgical incisions that have not fully healed prior to the first dose of the drug
11. patients with clinical cardiac symptoms or disease that are not well controlled, such as (1) NYHA class 2 or higher heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
12. subjects with active infection or unexplained fever >38.5 degrees during screening and prior to the first dose (subjects with fever arising from tumors may be enrolled, as determined by the investigator)
13. patients with a history of prior and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severely impaired lung function
14. live vaccines administered less than 4 weeks prior to study drug administration or likely to be administered during the study period
15. subjects with a known history of psychotropic substance abuse, alcoholism, or drug use
16. women who are pregnant or breastfeeding;
17. are of childbearing potential but unwilling to accept effective contraception
18. subjects who, in the opinion of the investigator, should be excluded from this study, for example, subjects who, in the judgment of the investigator, have other factors that might force the study to be terminated mid-study, such as, other serious illnesses (including psychiatric illnesses) requiring comorbid treatment, serious laboratory test abnormalities, accompanying family or social factors that would compromise the safety of the subject, or data and sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | through disease progression, an average of 6 months
  Proportion of patients whose tumors shrink by a certain amount and remain for a certain period of time

SECONDARY OUTCOMES:
DoR | through disease progression, an average of 6 months
  The time from the first evaluation of the tumor as CR or PR to the first evaluation of PD (Progressive Disease) or death from any cause
DCR | through disease progression, an average of 6 months
  Time from the start of the first evaluation of the tumor as CR, PR or SD to the first evaluation of PD (Progressive Disease) or death from any cause
PFS | through disease progression, an average of 1 6 months
  Time from treatment initiation to first tumor progression or death
OS | through patient death, an average of 1 year
  Time from the start of treatment to death from any cause